CLINICAL TRIAL: NCT05793970
Title: Evaluation of IL-6 Levels on Umbilical Cord
Brief Title: IL6 on Umbilical Cord (Evaluation of IL-6 Levels on Umbilical Cord)
Acronym: INFIL-6
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parma University Hospital (Other)
Responsible Party: Principal Investigator, Tullio Ghi, Full Professor, Parma University Hospital
Other Study IDs: 561/2021/OSS/AOUPR
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Intrauterine Infection; Fetus Disorder
MeSH Terms: conditions — Fetal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5mL of umbilical cord blood will be sampled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fetal inflammatory response syndrome (FIRS) is a major cause of non-hypoxic fetal intrapartum injury. One of the most common determinants of FIRS during labor is the exposure to an ongoing intra-amniotic infectious agent as in the event of a chorioamnionitis. Interleuchine-6 (IL-6) is considered a reliable hallmark of FIRS. No specific fetal heart rate pattern for the diagnosis of FIRS have been described so far at intrapartum Cardiotocography (CTG). The aim the present study is to investigate the correlation between intrapartum CTG findings and IL-6 levels on the arterial cord.

DETAILED DESCRIPTION:
The labor will be managed according to the local protocol and 5mL of blood will collected from the umbilical artery soon after birth to determine the IL-6 values. CardioTocography (CTG) traces will be retrospectively reviewed by two expert operators that will be blinded to the IL-6 results and will categorize them as "inflammatory" or "not inflammatory".

Inflammatory pattern will be defined in presence of 1) inappropriately high FHR for the given gestational age and/or 2) an increase >10% compared with the FHR baseline values at admission without preceding deceleration with/without reduced variability or absent cycling.

The association between CTG findings as the umbilical levels of IL6 will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies at term submitted to a continuous CTG tracing during labor

Exclusion Criteria:elective Cesarean Delivery, maternal tachycardia or pyrexia >38°C, drugs assumption

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: singleton pregnancies at term submitted to a continuous CTG tracing during labor
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-03-23 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
IL6 Levels | IL6 will be measured on the umbilical blood sampled within 5 minutes after birth
  correlation between intrapartum CTG findings and IL-6 levels on the arterial cord

CONTACTS AND LOCATIONS:
Overall Officials: Tullio Ghi, Professor, Principal Investigator — University of Parma
Locations (2):
- Italy (2):
  - University Hospital of Parma, Parma
  - Fondazione Universitaria Policlinico Gemelli, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jung E, Romero R, Yeo L, Diaz-Primera R, Marin-Concha J, Para R, Lopez AM, Pacora P, Gomez-Lopez N, Yoon BH, Kim CJ, Berry SM, Hsu CD. The fetal inflammatory response syndrome: the origins of a concept, pathophysiology, diagnosis, and obstetrical implications. Semin Fetal Neonatal Med. 2020 Aug;25(4):101146. doi: 10.1016/j.siny.2020.101146. Epub 2020 Oct 23. PMID 33164775
- [Background] Gotsch F, Romero R, Kusanovic JP, Mazaki-Tovi S, Pineles BL, Erez O, Espinoza J, Hassan SS. The fetal inflammatory response syndrome. Clin Obstet Gynecol. 2007 Sep;50(3):652-83. doi: 10.1097/GRF.0b013e31811ebef6. PMID 17762416
- [Background] Romero R, Chaemsaithong P, Docheva N, Korzeniewski SJ, Tarca AL, Bhatti G, Xu Z, Kusanovic JP, Chaiyasit N, Dong Z, Yoon BH, Hassan SS, Chaiworapongsa T, Yeo L, Kim YM. Clinical chorioamnionitis at term V: umbilical cord plasma cytokine profile in the context of a systemic maternal inflammatory response. J Perinat Med. 2016 Jan;44(1):53-76. doi: 10.1515/jpm-2015-0121. PMID 26360486
- [Background] Ren J, Qiang Z, Li YY, Zhang JN. Biomarkers for a histological chorioamnionitis diagnosis in pregnant women with or without group B streptococcus infection: a case-control study. BMC Pregnancy Childbirth. 2021 Mar 25;21(1):250. doi: 10.1186/s12884-021-03731-7. PMID 33765949